CLINICAL TRIAL: NCT04908904
Title: Acute Effects of Cafestol on Glucose Metabolism in Subjects With Type-2-diabetes.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: cafestol.acute.t2d
Record Dates: First submitted 2021-05-27; First posted 2021-06-01 (Actual); Last update posted 2022-02-28 (Actual); Status verified 2021-05

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — cafestol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cafestol (Active Comparator): 12 mg cafestol
  Interventions: Dietary Supplement: Cafestol
- Placebo (Placebo Comparator): Placebo
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Cafestol — Capsule with 12 mg cafestol
  Arms: Cafestol
Dietary Supplement: Placebo — Placebo capsule without cafestol
  Arms: Placebo

SUMMARY:
Acute, double-blinded, randomized, cross-over cafestol intervention study with sixteen participants with T2D participating in two OGTTs.

DETAILED DESCRIPTION:
The study is an acute, double-blinded, randomized, cross-over intervention study with sixteen participants with T2D. Initially, a blood sample is obtained (t=-15 min) and at time point 0, the participants will ingest a tablet containing either 12 mg cafestol or placebo. Immediately hereafter an OGTT commences with ingestion of a 75 g glucose solution. In the following 3 hours blood samples are collected at time points 0, 15, 30, 60, 90, 120 and 180 min. The samples will be used for determination of plasma glucose, insulin and cafestol, as well as GLP-1 and GIP. After a one-week washout period, the subject will undergo the same set-up again, however now with the opposite intervention / placebo.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 Diabetes defined by standard Danish guidelines
* HbA1c ≥48 mmol/mol unless successfully treated with antidiabetic drugs and/or diet/exercise intervention

Exclusion Criteria:

* In treatment with insulin
* Pregnancy
* Planned pregnancy
* Breastfeeding
* Significant comorbidity expected to unable the subject from completing visits

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-05-27 (Actual); Primary Completion 2022-02-16 (Actual); Study Completion 2022-02-16 (Actual)

PRIMARY OUTCOMES:
Area under the curve for glucose | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for glucose during OGTT after ingestion of cafestol or placebo capsule

SECONDARY OUTCOMES:
Area under the curve for insulin-response | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for insulin response during OGTT after ingestion of cafestol or placebo capsule
Area under the curve for cafestol | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for cafestol during OGTT after ingestion of cafestol or placebo capsule
Area under the curve for GLP-1 | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for GLP-1 (glucagon-like peptide-1) during OGTT after ingestion of cafestol or placebo capsule
Area under the curve for GIP | -15 to 180 minutes from ingestion of intervention/placebo capsule and 75 g. glucose solution
  Area under the curve for GIP (Glucose-dependent insulinotropic polypeptide) during OGTT after ingestion of cafestol or placebo capsule

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Aarhus, Aarhus, Aarhus N, Denmark

IPD SHARING:
Plan to Share IPD: Undecided